CLINICAL TRIAL: NCT04749498
Title: Effects of Barley and Oat Breads on Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Zeynep Caferoglu, PhD, Assistant Professor Doctor, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: TSA-2019-8761
Record Dates: First submitted 2021-02-06; First posted 2021-02-11 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Healthy; Appetitive Behavior
Keywords: appetite; barley; β-glucan; bread; glucose; oats; food intake
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- White Bread (Active Comparator): White bread with a standard test breakfast
  Interventions: Other: White Bread
- Whole Wheat Bread (Active Comparator): Whole wheat bread with a standard test breakfast
  Interventions: Other: Whole Wheat Bread
- Barley Bread (Experimental): Barley bread with a standard test breakfast
  Interventions: Other: Barley Bread
- Oat Bread (Experimental): Oat bread with a standard test breakfast
  Interventions: Other: Oat Bread

INTERVENTIONS:
Other: White Bread — Test breakfast with white bread was served after 12-hours of fasting and participants were asked to consume the meal in full, within 15 minutes.
  Arms: White Bread
Other: Whole Wheat Bread — In a crossover design, this bread was served with a standard breakfast to compare other breads.
  Arms: Whole Wheat Bread
Other: Barley Bread — In a crossover design, this bread was served with a standard breakfast to compare other breads.
  Arms: Barley Bread
Other: Oat Bread — In a crossover design, this bread was served with a standard breakfast to compare other breads.
  Arms: Oat Bread

SUMMARY:
This study aimed to compare the postprandial effects of ß-glucan derived from oats bread (OB) and barley bread (BB) on appetite and glycemia. A randomized, double-blind, crossover trial included 20 healthy individuals. All participants consumed BB, white bread (WB), and whole wheat bread (WWB) with a standard breakfast and then were served an ad libitum lunch on four different days. A visual analog scale (VAS) was used to assess appetite before breakfast and at 15, 30, 60, 90, 120, 150, and 180 minutes after breakfast. Blood glucose levels were measured at 0, 15, 30, 45, 60, 90, and 120 minutes. Postprandial appetite and glucose responses were quantified as the incremental area under the curve (iAUC) calculated according to the trapezoidal rule.

DETAILED DESCRIPTION:
This study aimed to compare the postprandial effects of ß-glucan on glycemia and appetite of breads derived from oats and barley, which are the best natural grain sources. In addition, the positive health effects of ß-glucan were sought to be determined independent of total dietary fiber intake, using not only WB as the control food but also WWB, which has a dietary fiber content equal to that of breads containing ß-glucan. This study was planned as a multicenter, randomized, double-blind, and crossover. Twenty healthy adults (10 men, 10 women) between the ages of 19-35 years, with normal body weight (BMI 18.5-25 kg /m2) were included in the study. Participants were selected from among Erciyes University students and staff in accordance with the inclusion criteria. The eating behaviors of all participants were also evaluated using the Dutch Eating Behavior Questionnaire before starting the study. Since the total score obtained from this questionnaire >3.5 is considered as restrictive eating behavior, these individuals were not included in the study.

Participants were served barley bread (BB), oat bread (OB), and white bread (WB), and whole wheat bread (WWB) with a standard breakfast on four different days at least two days apart. Breads were prepared with similar amounts of energy, protein, fat, carbohydrate, and fiber (except WB). The test meal was served to the participants at 09:00 and they were asked to consume it within 15 minutes. A visual analog scale (VAS) was used to assess appetite before breakfast and at 15, 30, 60, 90, 120, 150, and 180 minutes after breakfast. Furthermore, the separate VAS components such as hunger, fullness, desire to eat, and prospective food consumption were combined to produce an additional measure termed 'composite appetite score'. For the postprandial glucose assessment, blood glucose measurements were made with the finger-tip glucometer at 0, 15, 30, 45, 60, 90, and 120 minutes. Postprandial appetite and glucose responses were quantified as the incremental area under the curve (iAUC) calculated according to the trapezoidal rule.

At the end of three hours, the ad libitum lunch was served to the participants as a buffet-style, and the energy and macronutrient intakes in this meal were determined. All foods (meatballs, tuna, sauce pasta, yogurt, salad, white bread, apple, banana, yogurt drink, fruit juice, and water) were weighed using a calibrated kitchen scale with an accuracy of ±1g before being served. At lunch, the participants were asked to consume the foods they wanted and continue eating until they felt completely full. After the participants completed their consumption, the remaining amounts were reweighed and the difference with the initial amounts was accepted as the amount consumed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Normal-weight (BMI 18.5-25 kg/m2)
* 19-35 years
* Having a <3.5 score on the Dutch Eating Behavior Questionnaire (considered as unrestrictive eating behavior)

Exclusion Criteria:

* Applying an energy-restricted diet in the last three months
* Having a change in body weight >5 kg in the last three months
* Vegans
* Having any chronic diseases such as diabetes, hypertension, etc.
* Physician-diagnosed medications or conditions that influence metabolism
* Having fasting glucose >100 mg/dl
* Smoking
* Exercising heavily
* Having chewing/swallowing difficulties or sensitivity/allergies to any food to be used in the study
* Lack of appetite
* Pregnant and lactating women
* Skipping breakfast meals

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Postprandial appetite response | Three hours postprandial period (from fasting to 180 minutes after the test breakfast)
  The separate visual analog scale factors like hunger, fullness, desiring for eat, and prospective food consumption were combined to produce an additional measure termed 'composite appetite score'. This average appetite score was computed for 0, 15, 30, 60, 90, 120, 150, and 180 minutes using the following equation: [(hunger + desire to eat + prospective food consumption + (100 - fullness)]/4 Total scale score changes in a range of 0-100. Higher values represent a worse outcome. Postprandial apetite response was quantified as incremental area under the curve (iAUC), which was calculated according to the trapezoidal rule by using composite appetite scores at time points 0, 15, 30, 60, 90, 120, 150, and 180 minutes. Higher values represent a worse outcome.
Postprandial glucose response | Two hours postprandial period (from fasting to 120 minutes after the test breakfast)
  Postprandial glucose response was quantified as incremental area under the curve (iAUC), which was calculated according to the trapezoidal rule by using serum glucose values at time points 0, 15, 30, 45, 60, 90, and 120 minutes. Higher values represent a worse outcome.
Subsequent energy consumption | Three hours after consuming the test breakfast (at 180 minutes)
  Energy intake at ad libitum lunch was calculated.

SECONDARY OUTCOMES:
Visual appeal of test bread | Immediately after consuming test meal (at 15 minutes)
  Palatability of test meals was measured by using a visual analog scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating. VAS ratings were measured by using a question "How is the visual appeal of test meal? (Good - Bad)" at time points 15 minutes (immediately after consuming test meal). Total scale score changes in a range of 0-100. Higher values represent a worse outcome.
Smell of test bread | Immediately after consuming test meal (at 15 minutes)
  Palatability of test meals was measured by using a visual analog scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating. VAS ratings were measured by using a question "How is the smell of test meal? (Good - Bad)" at time points 15 minutes (immediately after consuming test meal). Total scale score changes in a range of 0-100. Higher values represent a worse outcome.
Taste of test bread | Immediately after consuming test meal (at 15 minutes)
  Palatability of test meals was measured by using a visual analog scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating. VAS ratings were measured by using a question "How is the taste of test meal? (Good - Bad)" at time points 15 minutes (immediately after consuming test meal). Total scale score changes in a range of 0-100. Higher values represent a worse outcome.
Aftertaste of test bread | Immediately after consuming test meal (at 15 minutes)
  Palatability of test meals was measured by using a visual analog scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating. VAS ratings were measured by using a question "Is there any perceived taste in your mouth after test meal? (Much - None)" at time points 15 minutes (immediately after consuming test meal). Total scale score changes in a range of 0-100. Higher values represent a better outcome.
Palatability of test bread | Immediately after consuming test meal (at 15 minutes)
  Palatability of test meals was measured by using a visual analog scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating. VAS ratings were measured by using a question "How is the palatability of test meal? (Good - Bad)" at time points 15 minutes (immediately after consuming test meal). Total scale score changes in a range of 0-100. Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Caferoglu, PhD, Principal Investigator — Erciyes University Faculty of Health Sciences 38039 Kayseri / Turkey
Locations (1):
- Erciyes University Faculty of Health Sciences, Kayseri, Kayseri̇, Turkey (Türkiye)

REFERENCES:
- [Derived] Caferoglu Z, Aytekin Sahin G, Gonulalan Z, Hatipoglu N. Effects of whole-grain barley and oat beta-glucans on postprandial glycemia and appetite: a randomized controlled crossover trial. Food Funct. 2022 Oct 3;13(19):10225-10234. doi: 10.1039/d2fo01717b. PMID 36124913

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT04749498/Prot_SAP_000.pdf